CLINICAL TRIAL: NCT01533376
Title: Treatment of Port-wine Mark in Sturge-Weber Syndrome Using Topical Timolol
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Principal Investigator, Dr. Alex V. Levin, MD, MHSc, Chief, Pediatric Ophthalmology and Ocular Genetics, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AVL-SWS-TT4PWM
Record Dates: First submitted 2012-02-11; First posted 2012-02-15 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Sturge Weber Syndrome; Port-wine Mark
Keywords: Sturge Weber; SWS; Timolol; Port wine mark
MeSH Terms: conditions — Sturge-Weber Syndrome | interventions — Timolol

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Timolol (Experimental): Participants in this group will receive topical timolol
  Interventions: Drug: Timolol
- Placebo (Placebo Comparator): Participants in this group will receive Preservative free artificial tear gel.
  Interventions: Drug: Preservative free artificial tear gel.

INTERVENTIONS:
Drug: Timolol — 0.5% timolol maleate ophthalmic gel-forming solution applied once
  Other Names: Timoptic-XE
  Arms: Timolol
Drug: Preservative free artificial tear gel. — Preservative free artificial tear gel applied topically twice a day.
  Arms: Placebo

SUMMARY:
Primary Objective:

• To assess the possible utility of topical timolol in the management of port-wine mark (PWM) in Sturge-Weber syndrome in children.

DETAILED DESCRIPTION:
Port-wine mark (PWM) represents a congenital capillary malformation,characterized by dilation and malformation of dermal capillaries that lack endothelial proliferation. It is frequently seen in the facial distribution of the trigeminal nerve. PWM persists throughout life and involves ~0.3% of the population. Although PWMs are found in other circumstances, ~ 3% of patients with facial PWM are also afflicted with Sturge-Weber syndrome. PWMs are cosmetic entities that often have serious social consequences, producing psychological trauma to both children and their parents. PWM does not involute with time, and, if left untreated, can develop deep purple coloration, tissue hypertrophy, and nodularity.

Laser therapy, which selectively destroys specific targets within the skin, is currently the most commonly used approach for treating PWM, although complete blanching of the PWM after laser is rarely achieved for most patients, and only 10-45% of patients with Sturge-Weber have shown satisfactory outcomes. Complications of pulsed dye laser treatment for PWM include pyogenic granuloma, scabbing, cutaneous scarring, and permanent hypo/hyperpigmentation. Laser treatment is relatively contraindicated in children with darker skin coloration due to the resulting hypopigmentation which may be equally unsightly. Laser treatment causes substantial discomfort and pain to patients, and often requires general anesthesia in children. This is particularly true since earlier treatment in infancy is desirable and yields increased successful resolution of the PWM. The hypertrophic PWM in later years is resistant to any treatment. Recently, propranolol was reported to successfully treat capillary hemangioma in infants.13 While the mechanism by which beta blockade improves hemangioma is unclear, ß2-mediated vasoconstrictive effects and the ensuing apoptosis of capillary endothelial cells may contribute to the positive therapeutic results.

Oral application of propranolol can cause severe systemic complications, including bronchospasm, vasospasm, hypoglycemia, hypotension, severe bradycardia, heart block, and congestive heart failure. Topical timolol solution, a β-blocker, has shown a similar ability to reduce capillary hemangioma of eyelids with little or no systemic effects in a small pilot study. Similar to capillary hemangioma, which is a proliferative lesion characterized by increased endothelial cell turnover, PWM is a capillary malformation with abnormal endothelial cells and large surface area of dilated capillaries. Thus, both capillary hemangioma and PWM share the similar characteristic of abnormal capillary endothelial cells.

This pilot study is designed to explore the potential role of topical timolol in the management of PWM. As PWM is so frequently associated with Sturge-Weber syndrome, a disorder in which approximately 50% of patients will develop glaucoma, this study will be conducted in an ophthalmology setting.

This study will consist of two arms. One group will receive timolol and the second group a placebo preservative free artificial tear gel. The groups will be divided with a ratio of 1:1 and the Timolol group will be matched with the placebo group by PWM location, age and race.

Both medications are to be applied and rubbed in by fingertip to the treatment site twice a day for 6 months by subject's parents/guardian. (Treatment site: 1x1 cm at inferior edge of facial PWM)

Follow-up schedule: 1 week after treatment initiation and then every 2 months for a period of six months.

ELIGIBILITY:
Inclusion criteria:

* Age from 2 years to 10 years
* Port-Wine Mark
* English fluent and literate substitute decision maker
* Substitute decision maker vision sufficient to read informed consent document

Exclusion criteria:

* Active ocular infection (conjunctivitis, keratitis,)
* History of systemic conditions including hypo/hypertension, hypoglycemia, bradycardia, asthma or any contraindication to beta blocker use
* Unable to comply with required follow-up
* Substitute decision maker not English fluent or not literate
* Substitute decision maker unable to read consent document
* Patient already using systemic beta-blocker or beta-agonist (Patients already using topical beta-blocker for glaucoma will not be excluded from study).

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2012-02; Primary Completion 2019-01 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Appearance of Port-wine Mark at treatment site | 12 months
  Changes of color and size of PWM at treatment site will determine efficacy of the topical timolol.

CONTACTS AND LOCATIONS:
Overall Officials: Alex V Levin, MD, MHSc, Principal Investigator — Wills Eye Institute
Locations (1):
- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hennedige AA, Quaba AA, Al-Nakib K. Sturge-Weber syndrome and dermatomal facial port-wine stains: incidence, association with glaucoma, and pulsed tunable dye laser treatment effectiveness. Plast Reconstr Surg. 2008 Apr;121(4):1173-1180. doi: 10.1097/01.prs.0000304606.33897.71. PMID 18349634
- [Background] Jia W, Sun V, Tran N, Choi B, Liu SW, Mihm MC Jr, Phung TL, Nelson JS. Long-term blood vessel removal with combined laser and topical rapamycin antiangiogenic therapy: implications for effective port wine stain treatment. Lasers Surg Med. 2010 Feb;42(2):105-12. doi: 10.1002/lsm.20890. PMID 20166161
- [Background] Chiummariello S, Mezzana P, Fioramonti P, Onesti MG, Alfano C, Scuderi N. The use of laser and Varioscope in the management of hemangiomas and vascular malformations. Acta Chir Plast. 2006;48(1):20-5. PMID 16722347
- [Background] Li W, Yamada I, Masumoto K, Ueda Y, Hashimoto K. Photodynamic therapy with intradermal administration of 5-aminolevulinic acid for port-wine stains. J Dermatolog Treat. 2010 Jul;21(4):232-9. doi: 10.3109/09546630903159099. PMID 20509816
- [Background] Kautz G, Kautz I, Segal J, Zehren S. Treatment of resistant port wine stains (PWS) with pulsed dye laser and non-contact vacuum: a pilot study. Lasers Med Sci. 2010 Jul;25(4):525-9. doi: 10.1007/s10103-009-0727-7. Epub 2009 Dec 15. PMID 20013138
- [Background] Maruani A. [Sturge-Weber syndrome]. Presse Med. 2010 Apr;39(4):482-6. doi: 10.1016/j.lpm.2009.07.030. Epub 2010 Mar 10. French. PMID 20219318
- [Background] Onesti MG, Fioramonti P, Carella S, Spinelli G, Scuderi N. Surgical and laser treatment of Sturge-Weber syndrome. Aesthetic Plast Surg. 2009 Jul;33(4):666-8. doi: 10.1007/s00266-009-9327-y. Epub 2009 Mar 19. PMID 19296147
- [Background] Latkowski IT, Wysocki MS, Siewiera IP. [Own clinical experience in treatment of port-wine stain with KTP 532 nm laser]. Wiad Lek. 2005;58(7-8):391-6. Polish. PMID 16425790
- [Background] Li G, Lin T, Wu Q, Zhou Z, Gold MH. Clinical analysis of port wine stains treated by intense pulsed light. J Cosmet Laser Ther. 2010 Feb;12(1):2-6. doi: 10.3109/14764170903449778. PMID 20085450
- [Background] Wareham WJ, Cole RP, Royston SL, Wright PA. Adverse effects reported in pulsed dye laser treatment for port wine stains. Lasers Med Sci. 2009 Mar;24(2):241-6. doi: 10.1007/s10103-008-0560-4. Epub 2008 Apr 17. PMID 18418641
- [Background] Minkis K, Geronemus RG, Hale EK. Port wine stain progression: a potential consequence of delayed and inadequate treatment? Lasers Surg Med. 2009 Aug;41(6):423-6. doi: 10.1002/lsm.20788. PMID 19588535
- [Background] Izikson L, Nelson JS, Anderson RR. Treatment of hypertrophic and resistant port wine stains with a 755 nm laser: a case series of 20 patients. Lasers Surg Med. 2009 Aug;41(6):427-32. doi: 10.1002/lsm.20793. PMID 19588532
- [Background] Leaute-Labreze C, Dumas de la Roque E, Hubiche T, Boralevi F, Thambo JB, Taieb A. Propranolol for severe hemangiomas of infancy. N Engl J Med. 2008 Jun 12;358(24):2649-51. doi: 10.1056/NEJMc0708819. No abstract available. PMID 18550886
- [Background] Siegfried EC, Keenan WJ, Al-Jureidini S. More on propranolol for hemangiomas of infancy. N Engl J Med. 2008 Dec 25;359(26):2846; author reply 2846-7. doi: 10.1056/NEJMc086443. No abstract available. PMID 19109584
- [Background] Guo S, Ni N. Topical treatment for capillary hemangioma of the eyelid using beta-blocker solution. Arch Ophthalmol. 2010 Feb;128(2):255-6. doi: 10.1001/archophthalmol.2009.370. No abstract available. PMID 20142555